CLINICAL TRIAL: NCT04264013
Title: Eggs as Nutrient-Rich Source of Protein to Enhance Activity-Related Health in Older Persons: The Eggs and actiVity in hEalth agiNg Pilot (EVEN-P) Trial
Brief Title: The Eggs and actiVity in hEalth agiNg Pilot (EVEN-P) Trial in Older Persons
Acronym: EVEN-P
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 7919
Record Dates: First submitted 2020-02-05; First posted 2020-02-11 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2022-04

CONDITIONS: Aging
Keywords: Muscle; Diet; Sarcopenia; Vascular health
MeSH Terms: conditions — Sarcopenia | interventions — Exercise; Diet; Eggs

STUDY DESIGN:
Intervention Model Description: The study will be a randomized parallel-group trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Placebo Comparator): Exercise
  Interventions: Behavioral: Exercise
- Exercise + Diet (Active Comparator): Exercise + eggs
  Interventions: Behavioral: Exercise plus diet (egg)

INTERVENTIONS:
Behavioral: Exercise — Participants will exercise in a supervised facility twice weekly and consume their habitual diet.
  Arms: Exercise
Behavioral: Exercise plus diet (egg) — Participants will exercise in a supervised facility twice weekly and consume an addiitonal 4 eggs per day.
  Arms: Exercise + Diet

SUMMARY:
Two of the most effective lifestyle-based approaches to reduce the risk of adverse health events and enhance quality of life with aging are exercise and a healthy diet. Currently, the Canadian recommended dietary allowance (RDA) for protein is 0.8 g/kg/day, however, several expert groups have advocated for a higher RDA of protein (~1.2 g/kg/day), along with more evenly distributed daily consumption, in older persons. Eggs are considered a nutrient-rich protein source but have recently been scrutinized. This study will compare a high-protein, egg-containing diet and a high-protein, non-egg diet in healthy older persons.

DETAILED DESCRIPTION:
This study will examine the impacts of an egg-containing diet and a non-egg diet in healthy older persons. Briefly, participants (healthy persons, age 60-75 years old) will consume their normal diet or their normal diet plus 4 eggs completing a structured exercise program (designed to meet Canada's Physical Activity Guidelines) for a total of 12 weeks. Participants will be randomly assigned to the Egg or Control (non-egg) group. Before and after the 12-week intervention, participants' undergo assessments of diet-quality, muscle health, fitness, bone health, and vascular health.

ELIGIBILITY:
Exclusion Criteria:

1. Use assistive walking devices (e.g. cane or walker)
2. Consume any analgesic (pain-relieving) or anti-inflammatory drug(s), prescription or non-prescription, chronically
3. A history of neuromuscular problems or muscle-wasting diseases
4. Any acute chronic illness, cardiac, pulmonary, liver, or kidney abnormalities, uncontrolled hypertension, insulin or non-insulin dependent diabetes or other metabolic disorders- all ascertained through medical screening questionnaires
5. Chronic consumption of statins (particularly simvastatin/Zocor and atorvastatin/Lipitor) used to lower cholesterol
6. Be on any medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories, or prescription-strength acne medications)
7. Have allergies or are not willing to consume eggs
8. Consume a vegetarian diet
9. Had significant weight gain or loss in the past 6 months
10. Have injuries preventing the safe completion of the exercise

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Dietary protein intake. | Pre- and post-intervention over 12 weeks
  Dietary protein intake (specifically meal-to-meal distribution) will be measured in all participants using a 3-day food log.

SECONDARY OUTCOMES:
Change in lean mass | Pre- and post-intervention over 12 weeks
  Composition by DXA
Strength | Pre- and post-intervention over 12 weeks
  Handgrip strength
Vascular health | Pre- and post-intervention over 12 weeks
  Measures of arterial compliance
Change in body fat mass | Pre- and post-intervention over 12 weeks
  Composition by DXA

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Phillips, Ph.D., Principal Investigator — McMaster University
Locations (1):
- Ivor Wynne Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No